CLINICAL TRIAL: NCT03508011
Title: A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of IMP4297 in Patients With Advanced Solid Tumors
Brief Title: A Study of IMP4297 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP4297-2016-CN01
Record Dates: First submitted 2018-01-08; First posted 2018-04-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumours; Breast Cancer; Ovarian Cancer; Prostate Cancer
Keywords: Breast Cancer; Ovarian Cancer; Prostate Cancer; Advanced solid tumours
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms | interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMP4297 (Experimental)
  Interventions: Drug: IMP4297

INTERVENTIONS:
Drug: IMP4297 — The dose levels will be escalated following a modified 3+3 dose escalation scheme.

SUMMARY:
This is a Phase I, first-in-human, open-label, dose-escalation study of IMP4297 administered orally once every day to patients with advanced solid tumors for whom standard therapy either does not exist or has proven to be ineffective or intolerable. Patients with advanced breast cancer, ovarian cancer or prostate cancer are preferred. There are two stages to this study: a dose-escalation stage and a dose-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. 18 Years to 70 Years (including 18 and 75 years)
3. Histologically or cytologically documented disease; incurable, advanced solid malignancy that has progressed on, or failed to respond to, at least one prior systemic therapy
4. Eastern Cooperative Oncology Group performance status of 0 or 1
5. In the dose expansion stage, patients with BRCA (breast carcinoma) mutation will be enrolled. Patients with breast cancer, ovarian cancer and prostate cancer are preferred.
6. In the dose escalation phase, at least one assessable lesion according to the RECIST 1.1 standard; In the dose expansion phase, at least one measurable lesion according to RECIST 1.1.

Exclusion Criteria:

1. Inadequate hematologic and organ function, defined by the following (hematologic parameters must be assessed ≥14 days after a prior treatment, if any):

   1. Absolute neutrophil count <1500 cells/µL
   2. Hemoglobin < 9 g/dL
   3. Total bilirubin > 1.5 × the upper limit of normal (ULN), with documented liver metastases total bilirubin > 3 × the ULN.
   4. Aspartate transaminase (AST) and/or alanine transaminase (ALT) > 2.5 × the ULN, with documented liver metastases AST and/or ALT levels > 5 × the ULN.
   5. Serum creatinine > 1.5 × the ULN, or creatinine clearance < 45 mL/min based on a documented 24-hour urine collection or Cockcroft-Gault calculation of glomerular filtration rate.
   6. International normalized ratio (INR) > 1.5 × the ULN or activated partial thromboplastin time (aPTT) > 1.5 × the ULN.

   The INR applies only to patients who do not receive therapeutic anti-coagulation.
2. Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, radiotherapy within 4 weeks prior to initiation of study treatment with the following exceptions:

   1. Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists for prostate cancer.
   2. Hormone-replacement therapy or oral contraceptives.
   3. Palliative radiation to bone metastases > 2 weeks prior to Day 1.
3. Adverse events from prior anti-cancer therapy that have not resolved to NCI CTCAE Grade ≤ 1, except for alopecia.
4. Prior therapies targeting PARP (poly-ADP ribose polymerase).
5. Clinical significant active infection
6. Known clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
7. Known human immunodeficiency virus infection
8. New York Heart Association Class II or greater congestive heart failure; history of myocardial infarction or unstable angina within 6 months prior to Day 1; history of stroke or transient ischemic attack within 6 months prior to Day 1
9. Active or untreated brain metastasis
10. Pregnant (positive pregnancy test) or lactating women
11. Male or female patients of child-producing potential unwilling to use double barrier contraception: condoms, sponge, foams, jellies, diaphragm or intrauterine device, contraceptives (oral, injectable or parenteral), implanon, or other avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
12. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
13. Inability to comply with study and follow-up procedures
14. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 57 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
The AEs (adverse event) of single and multiple doses of IMP4297 administered to participants with advanced solid tumors. | Each visit after IMP4297 administrated (through study completion, an average of 10 months)
  Evaluate the TEAE (treatment-emergent adverse event) of IMP4297
The maximum tolerated dose (MTD) and evaluate the dose limiting toxicities (DLTs) of IMP4297 | Within 28 days after IMP4297 administrated
  Evaluate DLT and determine the MTD

SECONDARY OUTCOMES:
Area Under Curve [AUClast, AUCINF] | Within 7 days after firstly single dose administrated
Area Under Curve [AUClast, AUCINF] | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Maximum plasma concentration (Cmax) | Within 7 days after firstly single dose administrated
Maximum plasma concentration (Cmax) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Time at which Cmax occurred (Tmax) | Within 7 days after firstly single dose administrated
Time at which Cmax occurred (Tmax) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Trough Concentrations (Ctrough) | Within 7 days after firstly single dose administrated
Trough Concentrations (Ctrough) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Clearance (CL/F) | Within 7 days after firstly single dose administrated
Clearance (CL/F) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)
Volume of distribution (Vd/F) | Within 7 days after firstly single dose administrated
Volume of distribution (Vd/F) | Within 16 days after first dose administrated in multiple dose cycle 1 (total 21 days in one cycle)

CONTACTS AND LOCATIONS:
Overall Officials: BingHe Xu, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; JunNing Cao, Doctor, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao J, Guo H, Ji D, Shen W, Zhang S, Hsieh CY, Xiong Cai S, Edward Tian Y, Xu C, Zhang P, Xu B. Safety, Tolerability, and Pharmacokinetics of Senaparib, a Novel PARP1/2 Inhibitor, in Chinese Patients With Advanced Solid Tumors: A Phase I Trial. Oncologist. 2023 Dec 11;28(12):e1259-e1267. doi: 10.1093/oncolo/oyad163. PMID 37338150